CLINICAL TRIAL: NCT03813849
Title: Sonographic Detection of Remnants After Surgical Evacuation of Missed Abortion
Brief Title: Remnants of Conception After Suction Evacuation of Missed Abortion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Mervat Sheikhelarab Elsedeek Ibrahim Omran, professor of obstetrics and gynecology, University of Alexandria
Other Study IDs: 0409/016
Record Dates: First submitted 2018-04-09; First posted 2019-01-23 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Miscarriage
Keywords: remnants of conception
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Sonographic examination of uterus after surgical evacuation

SUMMARY:
All women admitted for surgical evacuation of missed abortion after failure of medical treatment from June 2016 underwent transvaginal sonography immediately after completion of the procedure as judged by the operator to ensure absence of remnants.

DETAILED DESCRIPTION:
Women indicated for surgical evacuation of missed abortion up to 12 weeks were included. Standard surgical evacuation of uterus by suction followed by sharp curettage under general anaesthesia were done for all cases. When the operator judged the procedure as complete, transvaginal sonography was done by dedicated sonographer using portable ultrasound machine in theatre. If remnants were detected the procedure was repeated till the cavity seen empty.

ELIGIBILITY:
Inclusion Criteria:

multiparous. have missed abortion up to 12 weeks gestational age by dating. failed medical evacuation. consented for the procedure.

Exclusion Criteria:

suspicion of sepsis. Suspected molar pregnancy. previous evacuation trial. abnormal uterus like fibroids.

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: multiparous women, aged 18 to 45 years with missed abortion up to 12 weeks gestational age, with normal uterus and without suspicion of sepsis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-06-10 (Actual); Primary Completion 2020-01-30 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
presence remnants of conception | immediately after the end of the procedure
  transvaginal sonographic detection

CONTACTS AND LOCATIONS:
Locations (1):
- Shatby maternity university hospital, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided